CLINICAL TRIAL: NCT03030417
Title: A Phase I Study of Indenoisoquinoline LMP744 in Adults With Relapsed Solid Tumors and Lymphomas
Brief Title: Indenoisoquinoline LMP744 in Adults With Relapsed Solid Tumors and Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alice Chen, M.D., Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 170045; 17-C-0045
Record Dates: First submitted 2017-01-24; First posted 2017-01-25 (Estimated); Results first posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Solid Tumors; Lymphoma
Keywords: Topoisomerase I Inhibitor; Epithelial-Mesenchymal Transition; Pharmacodynamics; DNA Damage; Pharmacokinetics
MeSH Terms: conditions — Lymphoma | interventions — 6-(3-(2-hydroxyethyl)amino-1-propyl)-5,6-dihydro-2,3-dimethoxy-8,9-methylenedioxy-5,11-dioxo-11H-indeno(1,2-)isoquinoline; Ondansetron; Olanzapine; Lorazepam; Atropine; atropine sulfate-diphenoxylate hydrochloride drug combination; Loperamide; Diphenhydramine; Steroids; Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm - LMP744 (NSC 706744) (Experimental): LMP744 (NSC 706744) will be administered intravenous (IV) over 1 hour on days 1-5 of each 28-day cycle.
  Interventions: Drug: LMP744; Other: Ondansetron; Other: Olanzapine; Other: Lorazepam; Other: Diphenoxylate hydrocholoride (HCL) + Atropine Sulfate; Other: Loperamide; Other: Diphenhydramine; Other: Steroid; Other: Epinephrine

INTERVENTIONS:
Drug: LMP744 — Indenoisoquinolines, such as LMP744, are potent inhibitors of the enzyme topoisomerase I (Top1). Top1 is necessary for transcription, replication, recombination, and the repair of double-strand deoxyribonucleic acid (DNA) breaks. It relaxes the supercoiled DNA by introducing a single-strand break, generating a free strand that rotates around the Top1-bound DNA complex. In the absence of external triggers, Top1-DNA cleavage complexes are generally short lived. Top1 inhibitors are potent anticancer agents because they stabilize the formation of the Top1-DNA cleavage complex in tumor cells, which induces DNA damage, delays DNA repair, and results in cell cycle arrest and apoptosis. LMP744 exhibited antitumor activity with lower toxicity than other agents in preclinical studies. Treatment of patients with LMP744 is expected to reduce tumor burden at doses that are well-tolerated.
  Other Names: NSC 706744
Other: Ondansetron — Anti-emetic for nausea or vomiting.
  Other Names: Zofran ODT; Zuplenz; Zofran
Other: Olanzapine — Persistent nausea or vomiting.
  Other Names: Zyprexa Relprevv; Zyprexa Zydis; Zyprexa
Other: Lorazepam — Persistent nausea or vomiting.
  Other Names: Lorazepam Intensol; Ativan
Other: Diphenoxylate hydrocholoride (HCL) + Atropine Sulfate — Diphenoxylate hydrocholoride (HCL) 2.5 mg + Atropine Sulfate 0.025 mg/tablet for diarrhea.
  Other Names: Lomocot; Lomotil; Lonox; Vi-Atro
Other: Loperamide — Antidiarrheal. 4mg by mouth (PO) after first unformed stool and 2mg PO every 2 hours as long as unformed stools continue. No more than 16mg during a 24-hour period.
  Other Names: Imodium A-d; Diamode; Anti-Diarrheal (loperamide)
Other: Diphenhydramine — Diphenhydramine 50 mg intravenous (IV) for allergic reaction.
  Other Names: Benadryl; Nytol; Banophen
Other: Steroid — For allergic reaction at discretion of principal investigator.
Other: Epinephrine — For allergic reaction at discretion of principal investigator.
  Other Names: Adrenaline

SUMMARY:
Background:

The new drug LMP744 (NSC 706744) damages deoxyribonucleic acid (DNA). This causes cell death. Researchers want to see if it can treat certain kinds of cancer. They want to understand how the drug works and how it affects the body.

Objective:

To test the safety of LMP744 and find out the dose of the drug that can be safely given to humans.

Eligibility:

Adults at least 18 years old who have metastatic solid tumors or lymphoma, which have progressed after other treatment.

Design:

Participants will be screened with:

* Vital signs taken
* Blood and urine tests
* Heart tests
* Scans or ultrasound

Some participants will have a tumor sample taken 2 times. A small piece of tumor is removed by a small needle. A scan or ultrasound will guide the process.

The study will be done in 28-day cycles.

Each cycle, participants will get the study drug in a vein for 60 minutes once a day for 5 days.

For day 1 of cycle 1, participants will be admitted to the clinic and have blood and urine taken several times.

At the beginning of each cycle, participants will have a clinic visit and repeat some screening tests. They will also do this twice in the middle of cycle 1 and once in the middle of cycle 2.

After participants stop taking the study drug, they will be followed for 30 days. They may give blood samples. They will be contacted by phone to see how they are doing....

DETAILED DESCRIPTION:
Background:

* Indenoisoquinolines are non-camptothecin inhibitors of topoisomerase 1 (top1) with improved characteristics over their predecessors. Indenoisoquinolines have better chemical stability, producing stable deoxyribonucleic acid (DNA)-top1 cleavage complexes, and exhibit a preference for unique DNA cleavage sites, compared with their camptothecin counterparts.
* They have demonstrated activity against camptothecin-resistant cell lines and produce DNA-protein crosslinks, which are resistant to reversal. They also show less or no resistance to cells overexpressing the ATP-binding cassette (ABC) transporters, ATP-binding cassette super-family G member 2 (ABCG2), and multidrug resistance (MDR-1).

Primary Objectives:

-To establish the safety, tolerability and the maximum tolerated dose (MTD) of LMP744 (NSC 706744) administered intravenously (IV) daily for 5 days every day (QD) x 5) schedule in patients with refractory solid tumors and lymphomas.

Secondary Objectives:

-Characterize the pharmacokinetic (PK) profile of LMP744.

Exploratory Objectives:

* Evaluate the effect of LMP744 on markers of DNA damage phosphorylated H2AX (γH2AX), phosphorylated Nijmegen breakage syndrome 1 (pNbs1), pATR, excision repair cross-complementation group 1 (ERCC1), RAD51 recombinase (RAD51), Topo1cc, topoisomerase 1 (Top1), Schlafen family member 11 (SLFN11) and epithelial-mesenchymal transition (EMT) in circulating tumor cells (CTCs) and pre- and post- treatment tumor biopsies in patients at the expansion cohort.
* Assess preliminary antitumor activity of LMP744.
* Examine genomic alterations in circulating tumor DNA (ctDNA) that may be associated with response or resistance to treatment

Eligibility:

-Adult patients must have histologically documented, relapsed solid tumors which have progressed after one line of therapy, or lymphoma which has progressed after initial therapy and without potentially curative options, or patient refuses potentially curative therapy.

Study Design:

* Cycle 1 and subsequent cycles: Patients will receive LMP744 administered IV QD over 1 hour on days 1-5 followed by 23 days without drug (28-day cycle).
* Pharmacokinetic (PK) and pharmacodynamic (PD) samples will be collected. Tumor biopsies will be mandatory during the expansion phase.

LMP744 will be administered IV over 1 hour on days 1-5 of each 28-day cycle.

Blood samples for PK analyses will be collected at the following timepoints in cycle 1 only:

Day 1, prior to drug administration, 2 minutes (+/- 2 minutes) before end of infusion, and at appropriate time points post infusion (15 minutes, 30 minutes, and 1, 2, 4, and 6 hours post infusion)

Day 2, 24-hour (hr) post day 1 start of infusion (prior to day 2 infusion), and 2 minutes (+/- 2 minutes) before the end of infusion

Day 3, 24 hr post day 2 start of infusion (prior to day 3 infusion), and 2 minutes (+/- 2 minutes) before end of infusion

Day 4, 24 hr post day 3 start of infusion (prior to day 4 infusion), and 2 minutes (+/- 2 minutes) before end of infusion

Day 5, 24 hr post day 4 start of infusion (prior to day 5 infusion), and 2 minutes (+/- 2 minutes) before end of infusion

Day 8, 72 hr post day 5 start of infusion Blood for circulating tumor cells (CTCs) (optional) will be collected at baseline, on day 3 of

Cycle 1 (within 2 to 4 hours after the start of LMP744 infusion), on day 1 of every subsequent cycle (prior to drug infusion), and at disease progression.

Tumor biopsies (mandatory in expansion phase) will be obtained at baseline and then on day 2 (1-4 hours after the LMP744 infusion) in cycle 1 only.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Patients must have histologically documented metastatic solid tumors which have progressed after one line of therapy, or lymphoma which has progressed after initial therapy and without potentially curative options, or patient refuses potentially curative therapy.
  2. Patients must have measurable or evaluable disease
  3. Age greater than or equal to 18 years.
  4. Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
  5. Life expectancy of greater than 3 months.
  6. Patients must have normal organ and marrow function as defined below:

     leukocytes greater than or equal to 3,000/mcL

     absolute neutrophil count greater than or equal to 1,500/mcL

     platelets greater than or equal to 100,000/mcL

     total bilirubin within normal institutional limits

     Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT)/ alanine aminotransferase (ALT) serum glutamate-pyruvate transaminase (SGPT) less than or equal to 2.5 institutional upper limit of normal (ULN)

     Serum creatinine less than or equal to 1.5 institutional ULN

     OR

     creatinine clearance greater than or equal to 60 mL/min/1.73 m^2 for patients with serum creatinine levels greater than 1.5 x higher than institutional normal.
  7. Anticoagulation with low-molecular-weight heparin (LMWH) or any direct oral anticoagulant (direct oral anticoagulants (DOAC), e.g., rivaroxaban, apixaban, dabigatran, or edoxaban) will be permitted. Patients receiving treatment with warfarin will be given the option to switch to LMWH or a DOAC.
  8. Patients must have recovered to grade 1 or baseline from adverse events (AEs) and/or toxicity of prior chemotherapy or biologic therapy. They must not have had chemotherapy, biologic therapy, or definitive radiotherapy within 4 weeks (6 weeks for nitrosoureas and mitomycin C) or 5 half-lives, whichever is shorter, prior to entering the study. Palliative-intent radiotherapy (30 Gray (Gy) or less) must be completed at least 2 weeks prior to start of treatment and may not be to a lesion that is included as measurable disease. Patients must be greater than or equal to 2 weeks since any investigational agent administered as part of a Phase 0 study (where a sub-therapeutic dose of drug is administered) at the PI's discretion and should have recovered to grade 1 or baseline from any toxicities.
  9. Patients receiving denosumab or bisphosphonates for any cancer or undergoing androgen deprivation therapy for prostate cancer are eligible for this therapy.
  10. Prior therapy with topoisomerase I inhibitors is allowed.
  11. Patients with known human immunodeficiency virus (HIV)-positive status are eligible provided the following criteria are met: cluster of differentiation 4 (CD4) count >350/mm^3, an undetectable viral load, and not receiving prophylaxis antibiotics. Diagnostic HIV testing will not be performed during screening or throughout this study.
  12. The effects of LMP744 (NSC 706744) on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Women and men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of LMP744 administration.
  13. Ability to understand and the willingness to sign a written informed consent document.
  14. Willingness to provide blood and new tumor biopsy samples for research purposes if on the expansion phase of the study.

EXCLUSION CRITERIA:

1. Patients who are receiving any other investigational agents.
2. Patients with clinically significant illnesses which would compromise participation in the study, including, but not limited to active or uncontrolled infection, immune deficiencies, Hepatitis B, Hepatitis C, uncontrolled diabetes, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
3. Patients with known brain metastases or carcinomatous meningitis are excluded from this clinical trial, with the exception of patients whose brain metastatic disease status has remained stable for greater than or equal to 1 month after treatment of the brain metastases. Patients on anti-seizure medications or steroid therapy may be enrolled at the discretion of the Principal Investigator.
4. Pregnant women are excluded from this study because LMP744 is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with LMP744, breastfeeding should be discontinued if the mother is treated.

INCLUSION OF WOMEN AND MINORITIES:

Both men and women of all races and ethnic groups are eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice P Chen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. All collected IPD will be shared with collaborators under the terms of collaborative agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Requests for all collected individual participant data (IPD) data from clinical trials, conducted under a binding collaborative agreement between National Cancer Institute (NCI)/Division of Cancer Treatment and Diagnosis (DCTD) and a pharmaceutical/biotechnology company, that are not under Data and Safety Monitoring Board (DSMB) monitoring must be in compliance with the terms of the binding collaborative agreement and must be approved by NCI/DCTD and the Pharmaceutical Collaborator (i.e., the NCI Experimental Therapeutics Clinical Trials Network (ETCTN) Director in conjunction with the NCI/DCTD Regulatory Affairs Branch).

REFERENCES:
- [Background] Antony S, Kohlhagen G, Agama K, Jayaraman M, Cao S, Durrani FA, Rustum YM, Cushman M, Pommier Y. Cellular topoisomerase I inhibition and antiproliferative activity by MJ-III-65 (NSC 706744), an indenoisoquinoline topoisomerase I poison. Mol Pharmacol. 2005 Feb;67(2):523-30. doi: 10.1124/mol.104.003889. Epub 2004 Nov 5. PMID 15531731
- [Background] Antony S, Agama KK, Miao ZH, Takagi K, Wright MH, Robles AI, Varticovski L, Nagarajan M, Morrell A, Cushman M, Pommier Y. Novel indenoisoquinolines NSC 725776 and NSC 724998 produce persistent topoisomerase I cleavage complexes and overcome multidrug resistance. Cancer Res. 2007 Nov 1;67(21):10397-405. doi: 10.1158/0008-5472.CAN-07-0938. PMID 17974983
- [Background] Meng LH, Liao ZY, Pommier Y. Non-camptothecin DNA topoisomerase I inhibitors in cancer therapy. Curr Top Med Chem. 2003;3(3):305-20. doi: 10.2174/1568026033452546. PMID 12570765
- [Derived] O'Sullivan Coyne G, Kummar S, Rubinstein LV, Wilsker D, Moore N, Hogu M, Piekarz R, Covey J, Beumer JH, Ferry-Galow KV, Villaruz LC, Hollingshead MG, Holleran JL, Deppas JJ, Pommier Y, Ko B, Johnson BC, Parchhment RE, Ivy P, Doroshow JH, Chen AP. Phase 1 studies of the indenoisoquinolines LMP776 and LMP744 in patients with solid tumors and lymphomas. Cancer Chemother Pharmacol. 2025 May 29;95(1):58. doi: 10.1007/s00280-025-04778-5. PMID 40439882
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-C-0045.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Trmt) Assignment (Assign.) 1: LMP744 (MJ-III65 Hydrochloride) 6mg/m^2: Participants with metastatic solid tumors that have progressed after one line of therapy, or lymphoma that has progressed after all therapy. LMP744 (MJ-III65 hydrochloride) 6mg/m^2 intravenous over 1 hour on days 1-5 of each 28 day cycle.
- Treatment Assignment 2: LMP744 (MJ-III65 Hydrochloride) 12mg/m^2: Participants with metastatic solid tumors that have progressed after one line of therapy, or lymphoma that has progressed after all therapy. LMP744 (MJ-III65 hydrochloride) 12mg/m^2 intravenous over 1 hour on days 1-5 of each 28 day cycle.
- Treatment Assignment 3: LMP744 (MJ-III65 Hydrochloride) 24mg/m^2: Participants with metastatic solid tumors that have progressed after one line of therapy, or lymphoma that has progressed after all therapy. LMP744 (MJ-III65 hydrochloride) 24mg/m^2 intravenous over 1 hour on days 1-5 of each 28 day cycle.
- Treatment Assignment 4: LMP744 (MJ-III65 Hydrochloride) 48mg/m^2: Participants with metastatic solid tumors that have progressed after one line of therapy, or lymphoma that has progressed after all therapy. LMP744 (MJ-III65 hydrochloride) 48mg/m^2 intravenous over 1 hour on days 1-5 of each 28 day cycle.
- Treatment Assignment 5: LMP744 (MJ-III65 Hydrochloride) 96mg/m^2: Participants with metastatic solid tumors that have progressed after one line of therapy, or lymphoma that has progressed after all therapy. LMP744 (MJ-III65 hydrochloride) 96mg/m^2 intravenous over 1 hour on days 1-5 of each 28 day cycle.
- Treatment Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2: Participants with metastatic solid tumors that have progressed after one line of therapy, or lymphoma that has progressed after all therapy. LMP744 (MJ-III65 hydrochloride) 190mg/m^2 intravenous over 1 hour on days 1-5 of each 28 day cycle.
- Trmt Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 Followed by Trmt Assign. 5: 96mg/m^2: Participants with metastatic solid tumors that have progressed after one line of therapy, or lymphoma that has progressed after all therapy. LMP744 (MJ-III65 hydrochloride) 190mg/m^2 intravenous over 1 hour on days 1-5 followed by 96mg/m^2 intravenous over 1 hour on days 1-5 of each 28 day cycle.
- Trmt Assign. 6:LMP744 190mg/m^2 Foll. by Trmt Assign. 5: 96mg/m^2 Foll. by Trmt Assign. 4: 48mg/m^2: Participants with metastatic solid tumors that have progressed after one line of therapy, or lymphoma that has progressed after all therapy. LMP744 (MJ-III65 hydrochloride) 190mg/m^2 intravenous over 1 hour on days 1-5 followed by 96mg/m^2 intravenous over 1 hour on days 1-5 followed by 48mg/m^2 intravenous over 1 hour on days 1-5 of each 28 day cycle.
- Treatment Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2: Participants with metastatic solid tumors that have progressed after one line of therapy, or lymphoma that has progressed after all therapy. LMP744 (MJ-III65 hydrochloride) 260mg/m^2 intravenous over 1 hour on days 1-5 of each 28 day cycle.
- Trmt Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 Followed by Trmt Assign. 6: 190mg/m^2: Participants with metastatic solid tumors that have progressed after one line of therapy, or lymphoma that has progressed after all therapy. LMP744 (MJ-III65 hydrochloride) 260mg/m^2 intravenous over 1 hour on days 1-5 followed by 190mg/m^2 intravenous over 1 hour on days 1-5 of each 28 day cycle.
- Treatment Assignment 8: LMP744 (MJ-III65 Hydrochloride) 360mg/m^2: Participants with metastatic solid tumors that have progressed after one line of therapy, or lymphoma that has progressed after all therapy. LMP744 (MJ-III65 hydrochloride) 360mg/m^2 intravenous over 1 hour on days 1-5 of each 28 day cycle. No participants were enrolled in this group.
- Treatment Assignment 9: LMP744 (MJ-III65 Hydrochloride) 500mg/m^2: Participants with metastatic solid tumors that have progressed after one line of therapy, or lymphoma that has progressed after all therapy. LMP744 (MJ-III65 hydrochloride) 500mg/m^2 intravenous over 1 hour on days 1-5 of each 28 day cycle. No participants were enrolled in this group.
- Enrolled But Not Treated: Participant was enrolled but not treated.
Period: Dose Escalation
Arm/Group | Treatment (Trmt) Assignment (Assign.) 1: LMP744 (MJ-III65 Hydrochloride) 6mg/m^2 | Treatment Assignment 2: LMP744 (MJ-III65 Hydrochloride) 12mg/m^2 | Treatment Assignment 3: LMP744 (MJ-III65 Hydrochloride) 24mg/m^2 | Treatment Assignment 4: LMP744 (MJ-III65 Hydrochloride) 48mg/m^2 | Treatment Assignment 5: LMP744 (MJ-III65 Hydrochloride) 96mg/m^2 | Treatment Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 | Trmt Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 Followed by Trmt Assign. 5: 96mg/m^2 | Trmt Assign. 6:LMP744 190mg/m^2 Foll. by Trmt Assign. 5: 96mg/m^2 Foll. by Trmt Assign. 4: 48mg/m^2 | Treatment Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 | Trmt Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 Followed by Trmt Assign. 6: 190mg/m^2 | Treatment Assignment 8: LMP744 (MJ-III65 Hydrochloride) 360mg/m^2 | Treatment Assignment 9: LMP744 (MJ-III65 Hydrochloride) 500mg/m^2 | Enrolled But Not Treated
Started | 1 | 1 | 3 | 1 | 1 | 9 | 0 | 0 | 10 | 1 | 0 | 0 | 0
Restaging | 1 | 1 | 0 | 1 | 1 | 9 | 0 | 0 | 7 | 1 | 0 | 0 | 0
Pharmacokinetic Sampling | 1 | 1 | 3 | 1 | 1 | 9 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Tumor Biopsies | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 1 | 1 | 3 | 1 | 1 | 9 | 0 | 0 | 10 | 1 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Dose Expansion
Arm/Group | Treatment (Trmt) Assignment (Assign.) 1: LMP744 (MJ-III65 Hydrochloride) 6mg/m^2 | Treatment Assignment 2: LMP744 (MJ-III65 Hydrochloride) 12mg/m^2 | Treatment Assignment 3: LMP744 (MJ-III65 Hydrochloride) 24mg/m^2 | Treatment Assignment 4: LMP744 (MJ-III65 Hydrochloride) 48mg/m^2 | Treatment Assignment 5: LMP744 (MJ-III65 Hydrochloride) 96mg/m^2 | Treatment Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 | Trmt Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 Followed by Trmt Assign. 5: 96mg/m^2 | Trmt Assign. 6:LMP744 190mg/m^2 Foll. by Trmt Assign. 5: 96mg/m^2 Foll. by Trmt Assign. 4: 48mg/m^2 | Treatment Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 | Trmt Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 Followed by Trmt Assign. 6: 190mg/m^2 | Treatment Assignment 8: LMP744 (MJ-III65 Hydrochloride) 360mg/m^2 | Treatment Assignment 9: LMP744 (MJ-III65 Hydrochloride) 500mg/m^2 | Enrolled But Not Treated
Started | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 1 | 0 | 0 | 0 | 0 | 1
Restaging | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Pharmacokinetic Sampling | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumor Biopsies | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 1 | 0 | 0 | 0 | 0 | 1 (Only a pre-treatment baseline biopsy was collected.)
Completed | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Disease progression before treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: No participants were enrolled in treatment assignment group 8 and 9.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment (Trmt) Assignment (Assign.) 1: LMP744 (MJ-III65 Hydrochloride) 6mg/m^2 | Treatment Assignment 2: LMP744 (MJ-III65 Hydrochloride) 12mg/m^2 | Treatment Assignment 3: LMP744 (MJ-III65 Hydrochloride) 24mg/m^2 | Treatment Assignment 4: LMP744 (MJ-III65 Hydrochloride) 48mg/m^2 | Treatment Assignment 5: LMP744 (MJ-III65 Hydrochloride) 96mg/m^2 | Treatment Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 | Trmt Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 Followed by Trmt Assign. 5: 96mg/m^2 | Trmt Assign. 6:LMP744 190mg/m^2 Foll. by Trmt Assign. 5: 96mg/m^2 Foll. by Trmt Assign. 4: 48mg/m^2 | Treatment Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 | Trmt Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 Followed by Trmt Assign. 6: 190mg/m^2 | Enrolled But Not Treated | Total
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 14 | 2 | 1 | 10 | 1 | 1 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 2 | 0 | 1 | 7 | 2 | 1 | 6 | 0 | 1 | 21
  >=65 years | 0 | 1 | 1 | 1 | 0 | 7 | 0 | 0 | 4 | 1 | 0 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (0) | 79 (0) | 55.67 (8.96) | 81 (0) | 39 (0) | 62.57 (12.18) | 49 (19.8) | 46 (0) | 61.1 (8.96) | 72 (0) | 43 (0) | 60.03 (12.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 0 | 1 | 4 | 2 | 0 | 1 | 0 | 0 | 9
  Male | 1 | 1 | 2 | 1 | 0 | 10 | 0 | 1 | 9 | 1 | 1 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 4
  Not Hispanic or Latino | 1 | 1 | 3 | 1 | 0 | 12 | 1 | 1 | 10 | 1 | 1 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 6
  White | 1 | 1 | 3 | 0 | 1 | 11 | 2 | 1 | 7 | 1 | 1 | 29
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 3 | 1 | 1 | 14 | 2 | 1 | 10 | 1 | 1 | 36

OUTCOME MEASURES:

1. Primary Outcome: Dose Escalation Phase: Maximum Tolerated Dose (MTD) of LMP744 (NSC 706744)
Description: Maximum tolerated dose (MTD) of LMP744 administered intravenously (IV) daily for 5 days (QD x 5) schedule in participants with refractory solid tumors and lymphomas. The MTD is the dose level at which no more than 1 in 6 participants experience dose-limiting toxicity (DLT), and the dose below that at which ≥ 2 (of ≤ 6) participants have DLT as a result of the drug. A DLT is Grade ≥3 non-hematologic toxicity except Grade 3 fatigue lasting ≤ 7 days. Grade 4 hematological toxicity if it meets the following criteria: Lymphopenia (any grade) will not be considered dose limiting for all participants; Anemia: Grade 4 anemia will be considered dose limiting. Any neurotoxicity Grade ≥2 that is not reversible to a Grade ≤1 within 2 weeks. Any non-hematologic Grade 2 toxicity that does not resolve to Grade ≤1 or baseline within 14 days despite adequate treatment, except for alopecia.
Time Frame: Cycle 1 (28 days)
Population: A total of 27/27 participants were analyzed: 27/27 participants who received LMP744 in the Escalation phase were analyzed.
Measure: Number; unit: mg/m^2
Groups:
- All Participants: Dose Escalation: All participants who received LMP744 at Treatment Assignment 1 (6 mg/m^2), Treatment Assignment 2 (12 mg/m^2), Treatment Assignment 3 (24 mg/m^2), Treatment Assignment 4 (48 mg/m^2), Treatment Assignment 5 (96 mg/m^2), Treatment Assignment 6 (190 mg/m^2), n=9/14, Treatment Assignment 7 (260 mg/m^2), and Treatment Assignment 7 (260 mg/m^2) followed by Treatment Assignment 6 (190 mg/m^2) were assessed for dose-limiting toxicities.
Arm/Group | All Participants
Number analyzed (Participants) | 27
mg/m^2 | 190

2. Secondary Outcome: Dose Escalation & Dose Expansion Phase: Area Under the Plasma Concentration vs. Time Curve Extrapolated to Infinity (AUC(INF) of LMP744 (NSC 706744)
Description: AUC is a measure of the serum concentration of LMP744 over time. It is used to characterize drug absorption.
Time Frame: Day 1, prior to drug administration, 2 minutes before end of infusion; 15 minutes, 30 minutes, and 1, 2, 4, and 6 hours post infusion on Day 1 and prior to start of infusion on Day 2.
Population: A total of 20/36 participants were analyzed: samples from 20/36 participants who had blood collected for pharmacokinetic analyses were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL x h
Arm/Group | Treatment (Trmt) Assignment (Assign.) 1: LMP744 (MJ-III65 Hydrochloride) 6mg/m^2 | Treatment Assignment 2: LMP744 (MJ-III65 Hydrochloride) 12mg/m^2 | Treatment Assignment 3: LMP744 (MJ-III65 Hydrochloride) 24mg/m^2 | Treatment Assignment 4: LMP744 (MJ-III65 Hydrochloride) 48mg/m^2 | Treatment Assignment 5: LMP744 (MJ-III65 Hydrochloride) 96mg/m^2 | Treatment Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 | Trmt Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 Followed by Trmt Assign. 5: 96mg/m^2 | Trmt Assign. 6:LMP744 190mg/m^2 Foll. by Trmt Assign. 5: 96mg/m^2 Foll. by Trmt Assign. 4: 48mg/m^2 | Treatment Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 | Trmt Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 Followed by Trmt Assign. 6: 190mg/m^2
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 9 | 0 | 0 | 4 | 0
ng/mL x h | 37.1 | 50.7 | 198 (54) | 462 | 1858 | 5752 (5251) |  |  | 4928 (2174) |

3. Secondary Outcome: Dose Escalation & Dose Expansion Phase: Apparent Half-Life of LMP744 (NSC 706744)
Description: Plasma decay half-life is the time measured for the plasma concentration of the drug to decrease by one half.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Treatment (Trmt) Assignment (Assign.) 1: LMP744 (MJ-III65 Hydrochloride) 6mg/m^2 | Treatment Assignment 2: LMP744 (MJ-III65 Hydrochloride) 12mg/m^2 | Treatment Assignment 3: LMP744 (MJ-III65 Hydrochloride) 24mg/m^2 | Treatment Assignment 4: LMP744 (MJ-III65 Hydrochloride) 48mg/m^2 | Treatment Assignment 5: LMP744 (MJ-III65 Hydrochloride) 96mg/m^2 | Treatment Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 | Trmt Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 Followed by Trmt Assign. 5: 96mg/m^2 | Trmt Assign. 6:LMP744 190mg/m^2 Foll. by Trmt Assign. 5: 96mg/m^2 Foll. by Trmt Assign. 4: 48mg/m^2 | Treatment Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 | Trmt Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 Followed by Trmt Assign. 6: 190mg/m^2
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 8 | 0 | 0 | 4 | 0
Hours | 0.22 | 0.52 | 3.54 (0.91) | 4.66 | 16.2 | 12.59 (5.11) |  |  | 5.79 (3.30) |

4. Secondary Outcome: Dose Escalation & Dose Expansion Phase: Time to Maximum (Tmax) Concentration of LMP744 (NSC 706744)
Description: Time to maximum (Tmax) concentration of LMP744 (NSC 706744).
Time Frame: Day(D)1, prior to drug administration, 2 minutes (min) before end of infusion; 15 min., 30 min., and 1, 2, 4, and 6 hours (hr) post infusion on D1. 24 hrs post D2, 3, & 4 start of infusion & 2 min. before end of infusion. 72 hrs post D5 start of infusion.
Measure: Median (Full Range); unit: Hours
Arm/Group | Treatment (Trmt) Assignment (Assign.) 1: LMP744 (MJ-III65 Hydrochloride) 6mg/m^2 | Treatment Assignment 2: LMP744 (MJ-III65 Hydrochloride) 12mg/m^2 | Treatment Assignment 3: LMP744 (MJ-III65 Hydrochloride) 24mg/m^2 | Treatment Assignment 4: LMP744 (MJ-III65 Hydrochloride) 48mg/m^2 | Treatment Assignment 5: LMP744 (MJ-III65 Hydrochloride) 96mg/m^2 | Treatment Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 | Trmt Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 Followed by Trmt Assign. 5: 96mg/m^2 | Trmt Assign. 6:LMP744 190mg/m^2 Foll. by Trmt Assign. 5: 96mg/m^2 Foll. by Trmt Assign. 4: 48mg/m^2 | Treatment Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 | Trmt Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 Followed by Trmt Assign. 6: 190mg/m^2
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 14 | 2 | 1 | 10 | 1
Hours | 1.0 | 1.0 | 1.1 [1.0 to 2.8] | 1.0 | 1.0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 | 1.0 [1.0 to 1.5] | 1.0

5. Secondary Outcome: Dose Escalation & Dose Expansion Phase: Maximum Concentration of LMP744 (NSC 706744)
Description: To determine the maximum observed plasma concentration of LMP744, blood samples will be collected from participants and analyzed using a validated liquid chromatography-mass spectrometry (LC-MS) or liquid Chromatography with tandem mass spectrometry (LC-MS-MS) method and calculated by non-compartmental analysis.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment (Trmt) Assignment (Assign.) 1: LMP744 (MJ-III65 Hydrochloride) 6mg/m^2 | Treatment Assignment 2: LMP744 (MJ-III65 Hydrochloride) 12mg/m^2 | Treatment Assignment 3: LMP744 (MJ-III65 Hydrochloride) 24mg/m^2 | Treatment Assignment 4: LMP744 (MJ-III65 Hydrochloride) 48mg/m^2 | Treatment Assignment 5: LMP744 (MJ-III65 Hydrochloride) 96mg/m^2 | Treatment Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 | Trmt Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 Followed by Trmt Assign. 5: 96mg/m^2 | Trmt Assign. 6:LMP744 190mg/m^2 Foll. by Trmt Assign. 5: 96mg/m^2 Foll. by Trmt Assign. 4: 48mg/m^2 | Treatment Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 | Trmt Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 Followed by Trmt Assign. 6: 190mg/m^2
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 14 | 2 | 1 | 10 | 1
ng/mL | 48.4 | 69.6 | 78.1 (49.6) | 446 | 433.1 | 1735.4 (1188.9) | 861.0 (108.9) | 839.0 | 1560.9 (605.5) | 1160.1

6. Secondary Outcome: Dose Escalation & Dose Expansion Phase: Percent Change in End of Infusion Concentration of LMP744 (NSC 706744)
Description: Percent change in end of infusion drug concentration is a measure of LMP744 (NSC 706744) accumulation in the bloodstream from Day 1 to Day 5.
Time Frame: Day 1 at end of infusion to Day 5 end of infusion.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Treatment (Trmt) Assignment (Assign.) 1: LMP744 (MJ-III65 Hydrochloride) 6mg/m^2 | Treatment Assignment 2: LMP744 (MJ-III65 Hydrochloride) 12mg/m^2 | Treatment Assignment 3: LMP744 (MJ-III65 Hydrochloride) 24mg/m^2 | Treatment Assignment 4: LMP744 (MJ-III65 Hydrochloride) 48mg/m^2 | Treatment Assignment 5: LMP744 (MJ-III65 Hydrochloride) 96mg/m^2 | Treatment Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 | Trmt Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 Followed by Trmt Assign. 5: 96mg/m^2 | Trmt Assign. 6:LMP744 190mg/m^2 Foll. by Trmt Assign. 5: 96mg/m^2 Foll. by Trmt Assign. 4: 48mg/m^2 | Treatment Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 | Trmt Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 Followed by Trmt Assign. 6: 190mg/m^2
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 9 | 0 | 0 | 2 | 0
Percent change | 8.8 | 33.2 | 6.9 (35.6) | 20.1 | 41.6 | -14.1 (43.0) |  |  | 25.8 (10.4) |

7. Other Pre Specified Outcome: Dose Escalation & Dose Expansion Phase: Percentage of Participants With Confirmed Objective Response Following Treatment With LMP744 (NSC 706744)
Description: Antitumor activity is evaluated using the rate of confirmed objective responses according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria (i.e., at least a 30% decrease in the sum of the diameters of target lesions compared to the sum of baseline diameters).
Time Frame: Tumor re-staging was performed every 2 cycles for the first year on study then every 3 cycles thereafter until a participant met criteria to be removed from the study; a median of 2 cycles completed and a full range of 0-31 cycles completed.
Population: A total of 35/36 participants were analyzed: tumor measurements from 35/36 participants who had radiologic imaging were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment (Trmt) Assignment (Assign.) 1: LMP744 (MJ-III65 Hydrochloride) 6mg/m^2 | Treatment Assignment 2: LMP744 (MJ-III65 Hydrochloride) 12mg/m^2 | Treatment Assignment 3: LMP744 (MJ-III65 Hydrochloride) 24mg/m^2 | Treatment Assignment 4: LMP744 (MJ-III65 Hydrochloride) 48mg/m^2 | Treatment Assignment 5: LMP744 (MJ-III65 Hydrochloride) 96mg/m^2 | Treatment Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 | Trmt Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 Followed by Trmt Assign. 5: 96mg/m^2 | Trmt Assign. 6:LMP744 190mg/m^2 Foll. by Trmt Assign. 5: 96mg/m^2 Foll. by Trmt Assign. 4: 48mg/m^2 | Treatment Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 | Trmt Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 Followed by Trmt Assign. 6: 190mg/m^2
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 14 | 2 | 1 | 10 | 1
Percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 50 | 0 | 0 | 0

8. Other Pre Specified Outcome: Dose Expansion Phase: Percent of Nuclear Area Positive (NAP) for Phosphorylated Nibrin (pNbs1) Staining
Description: Levels of pNbs1 in paired pre-treatment and on-treatment tumor biopsies were quantified in response to treatment with LMP744 (NSC 706744)
Time Frame: Baseline (pre-treatment) and Cycle 1 Day 1 at 1-4 hours after the end of the LMP744 (NSC 706744) infusion.
Population: A total of 6/36 participants were analyzed: paired biopsy samples from 6 participants in the expansion phase were collected for pharmacodynamic analyses.
Measure: Mean (Standard Deviation); unit: Percent of Nuclear Positive Area (NAP)
Arm/Group | Treatment (Trmt) Assignment (Assign.) 1: LMP744 (MJ-III65 Hydrochloride) 6mg/m^2 | Treatment Assignment 2: LMP744 (MJ-III65 Hydrochloride) 12mg/m^2 | Treatment Assignment 3: LMP744 (MJ-III65 Hydrochloride) 24mg/m^2 | Treatment Assignment 4: LMP744 (MJ-III65 Hydrochloride) 48mg/m^2 | Treatment Assignment 5: LMP744 (MJ-III65 Hydrochloride) 96mg/m^2 | Treatment Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 | Trmt Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 Followed by Trmt Assign. 5: 96mg/m^2 | Trmt Assign. 6:LMP744 190mg/m^2 Foll. by Trmt Assign. 5: 96mg/m^2 Foll. by Trmt Assign. 4: 48mg/m^2 | Treatment Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 | Trmt Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 Followed by Trmt Assign. 6: 190mg/m^2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 0 | 0
Percent of Nuclear Positive Area (NAP)
  Pre-Treatment |  |  |  |  |  | 1.2 (0.7) | 0.2 (0.1) |  |  |
  On-Treatment (after end of infusion) |  |  |  |  |  | 1.5 (1.0) | 0.4 (0.2) |  |  |

9. Other Pre Specified Outcome: Dose Expansion Phase: Percent of Nuclear Area Positive (NAP) for RAD Recombinase (Rad51) Staining
Description: Levels of Rad51 in paired pre-treatment and on-treatment tumor biopsies were quantified in response to treatment with LMP744 (NSC 706744)
Time Frame: Baseline (pre-treatment) and Cycle 1 Day 1 at 1-4 hours after the end of the LMP744 (NSC 706744) infusion.
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percent of Nuclear Positive Area (NAP)
Arm/Group | Treatment (Trmt) Assignment (Assign.) 1: LMP744 (MJ-III65 Hydrochloride) 6mg/m^2 | Treatment Assignment 2: LMP744 (MJ-III65 Hydrochloride) 12mg/m^2 | Treatment Assignment 3: LMP744 (MJ-III65 Hydrochloride) 24mg/m^2 | Treatment Assignment 4: LMP744 (MJ-III65 Hydrochloride) 48mg/m^2 | Treatment Assignment 5: LMP744 (MJ-III65 Hydrochloride) 96mg/m^2 | Treatment Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 | Trmt Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 Followed by Trmt Assign. 5: 96mg/m^2 | Trmt Assign. 6:LMP744 190mg/m^2 Foll. by Trmt Assign. 5: 96mg/m^2 Foll. by Trmt Assign. 4: 48mg/m^2 | Treatment Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 | Trmt Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 Followed by Trmt Assign. 6: 190mg/m^2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 0 | 0
Percent of Nuclear Positive Area (NAP)
  Pre-Treatment |  |  |  |  |  | 0.2 (0.2) | 0.3 (0.1) |  |  |
  On-Treatment (after end of infusion) |  |  |  |  |  | 4.3 (2.6) | 3.4 (3.9) |  |  |

10. Other Pre Specified Outcome: Dose Expansion Phase: Percent of Nuclear Area Positive (NAP) for Topoisomerase I (Top1) Staining
Description: Levels of Top1 in paired pre-treatment and on-treatment tumor biopsies were quantified in response to treatment with LMP744 (NSC 706744)
Time Frame: Baseline (pre-treatment) and Cycle 1 Day 1 at 1-4 hours after the end of the LMP744 (NSC 706744) infusion.
Population: A total of 6/36 participants were analyzed: paired biopsy samples from 6 participants in the expansion phase were collected for pharmacodynamic analyses; one biopsy pair was not quantifiable.
Measure: Mean (Standard Deviation); unit: Percent of Nuclear Positive Area (NAP)
Arm/Group | Treatment (Trmt) Assignment (Assign.) 1: LMP744 (MJ-III65 Hydrochloride) 6mg/m^2 | Treatment Assignment 2: LMP744 (MJ-III65 Hydrochloride) 12mg/m^2 | Treatment Assignment 3: LMP744 (MJ-III65 Hydrochloride) 24mg/m^2 | Treatment Assignment 4: LMP744 (MJ-III65 Hydrochloride) 48mg/m^2 | Treatment Assignment 5: LMP744 (MJ-III65 Hydrochloride) 96mg/m^2 | Treatment Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 | Trmt Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 Followed by Trmt Assign. 5: 96mg/m^2 | Trmt Assign. 6:LMP744 190mg/m^2 Foll. by Trmt Assign. 5: 96mg/m^2 Foll. by Trmt Assign. 4: 48mg/m^2 | Treatment Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 | Trmt Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 Followed by Trmt Assign. 6: 190mg/m^2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0
Percent of Nuclear Positive Area (NAP)
  Pre-Treatment |  |  |  |  |  | 7.0 (3.7) | 2.2 (0.1) |  |  |
  On-Treatment (after end of infusion) |  |  |  |  |  | 6.4 (4.1) | 1.3 (1.3) |  |  |

11. Other Pre Specified Outcome: Dose Expansion Phase: Percent of Nuclear Area Positive (NAP) for Phosphorylated Krüppel Associated Box (KRAB) Domain-Associated Protein 1 (pKap1) Staining
Description: Levels of pKap1 in paired pre-treatment and on-treatment tumor biopsies were quantified in response to treatment with LMP744 (NSC 706744)
Time Frame: Baseline (pre-treatment) and Cycle 1 Day 1 at 1-4 hours after the end of the LMP744 (NSC 706744) infusion.
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percent of Nuclear Positive Area (NAP)
Units Other Than Participants: Samples
Arm/Group | Treatment (Trmt) Assignment (Assign.) 1: LMP744 (MJ-III65 Hydrochloride) 6mg/m^2 | Treatment Assignment 2: LMP744 (MJ-III65 Hydrochloride) 12mg/m^2 | Treatment Assignment 3: LMP744 (MJ-III65 Hydrochloride) 24mg/m^2 | Treatment Assignment 4: LMP744 (MJ-III65 Hydrochloride) 48mg/m^2 | Treatment Assignment 5: LMP744 (MJ-III65 Hydrochloride) 96mg/m^2 | Treatment Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 | Trmt Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 Followed by Trmt Assign. 5: 96mg/m^2 | Trmt Assign. 6:LMP744 190mg/m^2 Foll. by Trmt Assign. 5: 96mg/m^2 Foll. by Trmt Assign. 4: 48mg/m^2 | Treatment Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 | Trmt Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 Followed by Trmt Assign. 6: 190mg/m^2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 0 | 0
Number analyzed (Samples) | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 0 | 0
Percent of Nuclear Positive Area (NAP)
  Pre-Treatment |  |  |  |  |  | 0.3 (0.1) | 0.5 (NA) — There were 2 biopsy pairs analyzed, but only 1 was quantifiable, thus standard deviation cannot be determined. |  |  |
  On-Treatment (after end of infusion) |  |  |  |  |  | 0.2 (0.1) | 0.1 (0.2) |  |  |

12. Other Pre Specified Outcome: Dose Expansion Phase: Percent Change of Nuclei With ≥19 Topoisomerase 1 Cleavage Complex (Top1cc) Foci in Paired Biopsies
Description: Percent of nuclei with ≥19 Top1cc foci in paired pre-treatment and on-treatment tumor biopsies were quantified in response to treatment with LMP744 (NSC 706744)
Time Frame: Baseline (pre-treatment) and Cycle 1 Day 1 at 1-4 hours after the end of the LMP744 (NSC 706744) infusion.
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Treatment (Trmt) Assignment (Assign.) 1: LMP744 (MJ-III65 Hydrochloride) 6mg/m^2 | Treatment Assignment 2: LMP744 (MJ-III65 Hydrochloride) 12mg/m^2 | Treatment Assignment 3: LMP744 (MJ-III65 Hydrochloride) 24mg/m^2 | Treatment Assignment 4: LMP744 (MJ-III65 Hydrochloride) 48mg/m^2 | Treatment Assignment 5: LMP744 (MJ-III65 Hydrochloride) 96mg/m^2 | Treatment Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 | Trmt Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 Followed by Trmt Assign. 5: 96mg/m^2 | Trmt Assign. 6:LMP744 190mg/m^2 Foll. by Trmt Assign. 5: 96mg/m^2 Foll. by Trmt Assign. 4: 48mg/m^2 | Treatment Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 | Trmt Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 Followed by Trmt Assign. 6: 190mg/m^2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0
Percent change
  Pre-Treatment |  |  |  |  |  | 15.4 (14.0) | 7.6 (0.6) |  |  |
  On-Treatment (After end of infusion) |  |  |  |  |  | 13.3 (7.6) | 3.2 (4.4) |  |  |

13. Other Pre Specified Outcome: Dose Expansion Phase: Percent of Nuclear Area Positive (NAP) for Phosphorylated Form of Gamma H2A Histone Family Member X (γH2AX) Staining
Description: Levels of γH2AX in paired pre-treatment and on-treatment tumor biopsies were quantified in response to treatment with LMP744 (NSC 706744)
Time Frame: Baseline (pre-treatment) and Cycle 1 Day 1 at 1-4 hours after the end of the LMP744 (NSC 706744) infusion.
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percent of Nuclear Positive Area (NAP)
Arm/Group | Treatment (Trmt) Assignment (Assign.) 1: LMP744 (MJ-III65 Hydrochloride) 6mg/m^2 | Treatment Assignment 2: LMP744 (MJ-III65 Hydrochloride) 12mg/m^2 | Treatment Assignment 3: LMP744 (MJ-III65 Hydrochloride) 24mg/m^2 | Treatment Assignment 4: LMP744 (MJ-III65 Hydrochloride) 48mg/m^2 | Treatment Assignment 5: LMP744 (MJ-III65 Hydrochloride) 96mg/m^2 | Treatment Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 | Trmt Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 Followed by Trmt Assign. 5: 96mg/m^2 | Trmt Assign. 6:LMP744 190mg/m^2 Foll. by Trmt Assign. 5: 96mg/m^2 Foll. by Trmt Assign. 4: 48mg/m^2 | Treatment Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 | Trmt Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 Followed by Trmt Assign. 6: 190mg/m^2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 0 | 0
Percent of Nuclear Positive Area (NAP)
  Pre-Treatment |  |  |  |  |  | 0.5 (0.1) | 0.4 (0.0) |  |  |
  On-Treatment (after end of infusion) |  |  |  |  |  | 0.6 (0.3) | 5.5 (7.0) |  |  |

14. Other Pre Specified Outcome: Dose Escalation & Dose Expansion Phase: Number of Participants With Presence and/or Absence of Grade 2 or Higher Dose Limiting Toxicity (DLT)
Description: Toxicity was assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A DLT is Grade ≥3 non-hematologic toxicity except Grade 3 fatigue lasting ≤ 7 days. Grade 4 hematological toxicity if it meets the following criteria: Lymphopenia (any grade) will not be considered dose limiting for all participants; Anemia: Grade 4 anemia will be considered dose limiting. Any neurotoxicity Grade ≥2 that is not reversible to a Grade ≤1 within 2 weeks will be considered dose limiting. Any non-hematologic Grade 2 toxicity that does not resolve to Grade ≤1 or baseline within 14 days despite adequate treatment, except for alopecia. Grade 2 is moderate. Grade 3 is severe. Grade 4 is life-threatening. Grade 5 is death related to adverse event.
Time Frame: Cycle 1 (28 days)
Population: A total of 35/36 participants were analyzed: 35/36 participants who enrolled received at least 1 dose of LMP744 (NSC 706744) and were evaluable for toxicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Trmt) Assignment (Assign.) 1: LMP744 (MJ-III65 Hydrochloride) 6mg/m^2 | Treatment Assignment 2: LMP744 (MJ-III65 Hydrochloride) 12mg/m^2 | Treatment Assignment 3: LMP744 (MJ-III65 Hydrochloride) 24mg/m^2 | Treatment Assignment 4: LMP744 (MJ-III65 Hydrochloride) 48mg/m^2 | Treatment Assignment 5: LMP744 (MJ-III65 Hydrochloride) 96mg/m^2 | Treatment Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 | Trmt Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 Followed by Trmt Assign. 5: 96mg/m^2 | Trmt Assign. 6:LMP744 190mg/m^2 Foll. by Trmt Assign. 5: 96mg/m^2 Foll. by Trmt Assign. 4: 48mg/m^2 | Treatment Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 | Trmt Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 Followed by Trmt Assign. 6: 190mg/m^2
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 14 | 2 | 1 | 10 | 1
Participants
  Grade 2 DLT | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 DLT | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 0
  Grade 4 DLT | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 5 DLT | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

15. Other Pre Specified Outcome: Dose Escalation & Dose Expansion Phase: Number of Grades 2, 3, 4 and/or 5 Dose-limiting Toxicities (DLT) by Dose Level
Description: as for outcome 14
Time Frame: Cycle 1 (28 days)
Population: as for outcome 14
Measure: Number; unit: toxicities
Arm/Group | Treatment (Trmt) Assignment (Assign.) 1: LMP744 (MJ-III65 Hydrochloride) 6mg/m^2 | Treatment Assignment 2: LMP744 (MJ-III65 Hydrochloride) 12mg/m^2 | Treatment Assignment 3: LMP744 (MJ-III65 Hydrochloride) 24mg/m^2 | Treatment Assignment 4: LMP744 (MJ-III65 Hydrochloride) 48mg/m^2 | Treatment Assignment 5: LMP744 (MJ-III65 Hydrochloride) 96mg/m^2 | Treatment Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 | Trmt Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 Followed by Trmt Assign. 5: 96mg/m^2 | Trmt Assign. 6:LMP744 190mg/m^2 Foll. by Trmt Assign. 5: 96mg/m^2 Foll. by Trmt Assign. 4: 48mg/m^2 | Treatment Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 | Trmt Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 Followed by Trmt Assign. 6: 190mg/m^2
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 14 | 2 | 1 | 10 | 1
toxicities
  Grade 2 DLT - Weight loss | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 DLT - Hypokalemia | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 6 | 0
  Grade 3 DLT - Anemia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 5 DLT - Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

16. Other Pre Specified Outcome: Dose Escalation & Dose Expansion Phase: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: From first drug administration through 30 days after the last dose of study drug is administered, an average of 12.9 months.
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Trmt) Assignment (Assign.) 1: LMP744 (MJ-III65 Hydrochloride) 6mg/m^2 | Treatment Assignment 2: LMP744 (MJ-III65 Hydrochloride) 12mg/m^2 | Treatment Assignment 3: LMP744 (MJ-III65 Hydrochloride) 24mg/m^2 | Treatment Assignment 4: LMP744 (MJ-III65 Hydrochloride) 48mg/m^2 | Treatment Assignment 5: LMP744 (MJ-III65 Hydrochloride) 96mg/m^2 | Treatment Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 | Trmt Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 Followed by Trmt Assign. 5: 96mg/m^2 | Trmt Assign. 6:LMP744 190mg/m^2 Foll. by Trmt Assign. 5: 96mg/m^2 Foll. by Trmt Assign. 4: 48mg/m^2 | Treatment Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 | Trmt Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 Followed by Trmt Assign. 6: 190mg/m^2
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 14 | 2 | 1 | 10 | 1
Participants | 1 | 1 | 3 | 1 | 1 | 14 | 2 | 1 | 10 | 1

ADVERSE EVENTS:
Time Frame: From first drug administration through 30 days after the last dose of study drug is administered, an average of 12.9 months.
Arm/Group | Treatment (Trmt) Assignment (Assign.) 1: LMP744 (MJ-III65 Hydrochloride) 6mg/m^2 | Treatment Assignment 2: LMP744 (MJ-III65 Hydrochloride) 12mg/m^2 | Treatment Assignment 3: LMP744 (MJ-III65 Hydrochloride) 24mg/m^2 | Treatment Assignment 4: LMP744 (MJ-III65 Hydrochloride) 48mg/m^2 | Treatment Assignment 5: LMP744 (MJ-III65 Hydrochloride) 96mg/m^2 | Treatment Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 | Trmt Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 Followed by Trmt Assign. 5: 96mg/m^2 | Trmt Assign. 6:LMP744 190mg/m^2 Foll. by Trmt Assign. 5: 96mg/m^2 Foll. by Trmt Assign. 4: 48mg/m^2 | Treatment Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 | Trmt Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 Followed by Trmt Assign. 6: 190mg/m^2
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/1 | 1/3 | 0/1 | 1/1 | 0/14 | 0/2 | 0/1 | 3/10 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1 | 1/3 | 0/1 | 1/1 | 9/14 | 2/2 | 0/1 | 4/10 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 3/3 | 1/1 | 1/1 | 14/14 | 2/2 | 1/1 | 10/10 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Trmt) Assignment (Assign.) 1: LMP744 (MJ-III65 Hydrochloride) 6mg/m^2 (N=1) | Treatment Assignment 2: LMP744 (MJ-III65 Hydrochloride) 12mg/m^2 (N=1) | Treatment Assignment 3: LMP744 (MJ-III65 Hydrochloride) 24mg/m^2 (N=3) | Treatment Assignment 4: LMP744 (MJ-III65 Hydrochloride) 48mg/m^2 (N=1) | Treatment Assignment 5: LMP744 (MJ-III65 Hydrochloride) 96mg/m^2 (N=1) | Treatment Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 (N=14) | Trmt Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 Followed by Trmt Assign. 5: 96mg/m^2 (N=2) | Trmt Assign. 6:LMP744 190mg/m^2 Foll. by Trmt Assign. 5: 96mg/m^2 Foll. by Trmt Assign. 4: 48mg/m^2 (N=1) | Treatment Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 (N=10) | Trmt Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 Followed by Trmt Assign. 6: 190mg/m^2 (N=1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GGT increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Infections and infestations - Other, Bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Disease Progession (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritoneal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden death NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophageal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Trmt) Assignment (Assign.) 1: LMP744 (MJ-III65 Hydrochloride) 6mg/m^2 (N=1) | Treatment Assignment 2: LMP744 (MJ-III65 Hydrochloride) 12mg/m^2 (N=1) | Treatment Assignment 3: LMP744 (MJ-III65 Hydrochloride) 24mg/m^2 (N=3) | Treatment Assignment 4: LMP744 (MJ-III65 Hydrochloride) 48mg/m^2 (N=1) | Treatment Assignment 5: LMP744 (MJ-III65 Hydrochloride) 96mg/m^2 (N=1) | Treatment Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 (N=14) | Trmt Assignment 6: LMP744 (MJ-III65 Hydrochloride) 190mg/m^2 Followed by Trmt Assign. 5: 96mg/m^2 (N=2) | Trmt Assign. 6:LMP744 190mg/m^2 Foll. by Trmt Assign. 5: 96mg/m^2 Foll. by Trmt Assign. 4: 48mg/m^2 (N=1) | Treatment Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 (N=10) | Trmt Assignment 7: LMP744 (MJ-III65 Hydrochloride) 260mg/m^2 Followed by Trmt Assign. 6: 190mg/m^2 (N=1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 5 (8) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 5 (8) | 2 (4) | 0 (0) | 2 (3) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (4) | 10 (21) | 2 (8) | 0 (0) | 8 (16) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 6 (7) | 2 (2) | 0 (0) | 4 (4) | 1 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 7 (14) | 2 (3) | 0 (0) | 5 (5) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, blood bilirubin increased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 4 (7) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorders - Other, Left Ventricular wall hypokinesis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Concentration impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (10) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Creatinine increased (Investigations) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 6 (11) | 2 (5) | 0 (0) | 7 (8) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (10) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Endocrine disorders - Other, Hypothyroid (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endocrine disorders - Other, TSH decrease (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endocrine disorders - Other, TSH increased (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophageal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other, Ptosis-R side (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 8 (9) | 2 (4) | 0 (0) | 5 (5) | 1 (3)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
GGT increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 6 (16) | 2 (6) | 0 (0) | 2 (3) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Gastrointestinal disorders - Other, Abdominal cramping (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, Early satiety (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal disorders - Other, Hematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, LEFT SIDED PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (9) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 2 (4) | 0 (0) | 4 (4) | 1 (1)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 11 (20) | 2 (6) | 1 (1) | 8 (11) | 1 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (3) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 6 (18) | 1 (1) | 0 (0) | 7 (13) | 1 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 8 (19) | 0 (0) | 1 (1) | 6 (15) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (26) | 1 (2) | 0 (0) | 5 (5) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (28) | 1 (6) | 0 (0) | 6 (11) | 1 (4)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 10 (14) | 2 (8) | 0 (0) | 4 (13) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 7 (17) | 0 (0) | 0 (0) | 4 (5) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (2) | 0 (0) | 2 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, Bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Investigations - Other, Back Spasms (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Investigations - Other, Weight Loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Investigations - Other, Discoloration right toe nail (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Investigations - Other, Chloestatic Pruritus (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Investigations - Other, Eosinophilia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Investigations - Other, Generalized edema (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Investigations - Other, Hyponatremia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Investigations - Other, TSH increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Investigations - Other, INR increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (7) | 10 (21) | 2 (15) | 0 (0) | 8 (18) | 1 (2)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolism and nutrition disorders - Other, Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other, Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other, Hyperphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Metabolism and nutrition disorders - Other, Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Muscle Cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (22) | 1 (2) | 0 (0) | 4 (6) | 1 (4)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (13) | 2 (4) | 0 (0) | 4 (5) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 8 (20) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, Glucosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, P/C ratio inc (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Reproductive system and breast disorders - Other, Pulmonic Insufficiency (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Pulmonic insufficiency (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Discoloration R toe nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, possibly sunburn (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Folliculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Intercostal incisional hernia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Skin discoloration - Face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Rash Poss sunburn (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Superficial thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, Pain, biopsy site (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 7 (16) | 2 (6) | 1 (2) | 4 (4) | 1 (1)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (13) | 2 (2) | 0 (0) | 4 (6) | 1 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (14) | 2 (3) | 0 (0) | 3 (8) | 0 (0)
Cardiac disorders - Other, Pulmonic Insufficiency (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 4 (4) | 0 (0)
Lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
TSH increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glucosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Discoloration R toe (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-06): https://cdn.clinicaltrials.gov/large-docs/17/NCT03030417/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-06): https://cdn.clinicaltrials.gov/large-docs/17/NCT03030417/ICF_001.pdf